CLINICAL TRIAL: NCT04967118
Title: Neonatal Pain Management and Pain Monitoring Using New Methods: A Randomized Controlled Trial With Crossover Design
Brief Title: Neonatal Pain Management and Pain Monitoring Using New Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Anna-Kaija Palomaa, PhD researcher, University of Oulu
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 296/2018
Record Dates: First submitted 2021-03-17; First posted 2021-07-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pain, Acute; Procedural Pain; Infant
MeSH Terms: conditions — Acute Pain; Pain, Procedural | interventions — Kangaroo-Mother Care Method; Sound; Vibration; Glucose; Gurmarin protein, Gymnema sylvestre

STUDY DESIGN:
Intervention Model Description: A crossover design with each child as his or her own control will be used to minimize interchild variability. Order of interventions will be randomly assigned by computer-generated program.
Who Masked: Outcomes Assessor
Masking Description: Two research assistants (NICU nurses) who are blinded to the intervention condition (30% oral glucose and combination of 30% oral glucose and the mother's heartbeat intervention) will be perform calculation of infant PIPP-R and NIAPAS scores independently. Calculating NIAPAS scores will requires observation of the neonate's body, so during the skin-to-skin contact the intervention condition cannot be blinded. NIRS signals will be analyzed by researchers who are unaware of the nature of intervention and whether they are analyzing a noxious or non-noxious stimulation. To minimize observer bias, research assistants and researchers analyzing the NIRS signal will not be permitted to attend data collection sessions and will not share datasets or communicate with each other regarding the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skin-to-skin contact (Experimental): Neonates will be placed ventral skin-to-skin position with their mother at least thirty minutes prior the heel lance to give time to calm down following transfer. Skin-to-skin positioning will be taken account comfortable position as possible for mother and the baby, easy to access heel for blood sample and interference minimizing during video recording and continuous NIRS, ECG and oxygen saturation measurement. Skin-to-skin contact will be continued for approximately fifteen minutes after completion of blood sampling. In addition, the neonates will be given a 30% oral glucose solution two minutes prior the heel lance.
  Interventions: Behavioral: Skin-to-skin contact
- Mother's heartbeats as sound and vibration (Experimental): Neonates will be placed in an incubator or a cot, depending on their gestational age, and will be supported on side position by nest-shaped rolls according to department's normal practice. The platform on which the mother's heartbeat will be played will be placed under mattress of the incubator or crib. The playing of the mother's recorded heartbeats will be started thirty minutes prior the heel lance and will be continued during and fifteen minutes after the blood sampling. In addition, the neonates will be given a 30% oral glucose solution two minutes prior the heel lance.
  Interventions: Behavioral: Mother's heartbeats as sound and vibration
- 30% oral glucose (Active Comparator): Neonates will be placed on in an incubator or a cot, depending on their gestational age, and will be supported on side position by nest-shaped rolls according to department's normal practice. The neonates will be given a 30% oral glucose solution two minutes prior the heel lance
  Interventions: Drug: 30% oral glucose

INTERVENTIONS:
Behavioral: Skin-to-skin contact — Diaper clad baby will be placed ventral position on bare chest of mother 30 minute prior to the heel lance
  Other Names: Kangaroo Mother Care
  Arms: Skin-to-skin contact
Behavioral: Mother's heartbeats as sound and vibration — The mother's heartbeat will be recorded and the heartbeat sounds will be saved to the platform. The platform will be placed under the infant's mattress and the heartbeat will be started 30 minute prior to the heel lance.
  Arms: Mother's heartbeats as sound and vibration
Drug: 30% oral glucose — The infant will be given 30% oral glucose solution 2 minutes before the injection
  Other Names: Sweet taste
  Arms: 30% oral glucose

SUMMARY:
The aim of this randomized controlled study with crossover design is to examine the effectiveness of mother-driven interventions, skin-to-skin contact (SSC) and recorded mother's heartbeats as sound and vibration (MHB), compared to oral glucose in relieving neonatal acute pain related to heel lance as a painful procedure.

The effectiveness of interventions will be assessed using validated pain scales (PIPP-R and NIAPAS), changes in sensory cortex activation (near-infrared spectroscopy, NIRS) and changes in physiological indicators (oxygen saturation, heart rate, respiratory rate). The secondary objectives will include evaluating the effectiveness of interventions in relation to infant recovery and evaluating the use of NIRS monitoring in relation to neonatal pain assessment scales.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age (GA) at birth 32+0 - 42+0
* Admitted to NICU
* Parents are able to read, write and speak Finnish

Exclusion Criteria:

* With a postnatal age of 14 days or more
* Apgar points were 6 or less at 5 minutes of age
* Has been found grade III or IV cerebral haemorrhage
* Major congenital anomalies
* Has intubated or receiving a nCPAP
* Has received analgesics or sedatives for less than 24 hours prior to the study

Ages: 32 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in scores of Premature Infant Pain profile-Revised (PIPP-R) scale | Baseline 1, measured pre-intervention
  Pain intensity will be assessed using pain assessment tool, the Premature Infant Pain Profile Revised (PIPP-R). PIPP-R is an internationally widely used multidimensional pain assessment scale consisting of three behavioral indicators, two physiological indicators, and two contextual indicators.
Change in scores of Premature Infant Pain profile-Revised (PIPP-R) scale | Baseline 2, measured pre-procedure
  Pain intensity will be assessed using pain assessment tool, the Premature Infant Pain Profile Revised (PIPP-R). PIPP-R is an internationally widely used multidimensional pain assessment scale consisting of three behavioral indicators, two physiological indicators, and two contextual indicators.
Change in scores of Premature Infant Pain profile-Revised (PIPP-R) scale | Measured during painful procedure
  Pain intensity will be assessed using pain assessment tool, the Premature Infant Pain Profile Revised (PIPP-R). PIPP-R is an internationally widely used multidimensional pain assessment scale consisting of three behavioral indicators, two physiological indicators, and two contextual indicators.
Change in scores of Premature Infant Pain profile-Revised (PIPP-R) scale | Measured immediately after painful procedure
  Pain intensity will be assessed using pain assessment tool, the Premature Infant Pain Profile Revised (PIPP-R). PIPP-R is an internationally widely used multidimensional pain assessment scale consisting of three behavioral indicators, two physiological indicators, and two contextual indicators.
Change in scores of Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | Baseline 1, measured pre-intervention
  Pain intensity will be assessed using pain assessment tool, the Neonatal Infant Acute Pain Assessment Scale (NIAPAS). NIAPAS is multidimensional pain assessment scale used in Finland. It consist of five behavioral indicators, three physiological indicators, and one contextual indicator.
Change in scores of Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | Baseline 2, measured pre-procedure
  Pain intensity will be assessed using pain assessment tool, the Neonatal Infant Acute Pain Assessment Scale (NIAPAS). NIAPAS is multidimensional pain assessment scale used in Finland. It consist of five behavioral indicators, three physiological indicators, and one contextual indicator.
Change in scores of Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | Measured during painful procedure
  Pain intensity will be assessed using pain assessment tool, the Neonatal Infant Acute Pain Assessment Scale (NIAPAS). NIAPAS is multidimensional pain assessment scale used in Finland. It consist of five behavioral indicators, three physiological indicators, and one contextual indicator.
Change in scores of Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | Measured immediately after painful procedure
  Pain intensity will be assessed using pain assessment tool, the Neonatal Infant Acute Pain Assessment Scale (NIAPAS). NIAPAS is multidimensional pain assessment scale used in Finland. It consist of five behavioral indicators, three physiological indicators, and one contextual indicator.
Change in the activation in the somatosensory cortical areas following the noxious stimulation (baseline) | Baseline 1, measured pre-intervention
  In this study pain will be assessed measuring changes cortical hemodynamics by near-infrared spectroscopy (NIRS). A 2-channel NIRS will be used. The emitted probe provides near-infrared light through on optical fiber will be is placed slightly posterior to Cz position with reference to the international EEG 10-20 system. The receive probes will be fastened over somatosensory and occipital area. In the area of the somatosensory cortex, receive probes will be placed 2 to 4 cm from the emitted probe so that they are placed slightly behind C3 or C4 point. The occipital region receive probe will be attached 2 to 4 cm from the emitted probe.
Change in the activation in the somatosensory cortical areas following the noxious stimulation | Baseline 2, measured pre-procedure
  In this study pain will be assessed measuring changes cortical hemodynamics by near-infrared spectroscopy (NIRS). A 2-channel NIRS will be used. The emitted probe provides near-infrared light through on optical fiber will be is placed slightly posterior to Cz position with reference to the international EEG 10-20 system. The receive probes will be fastened over somatosensory and occipital area. In the area of the somatosensory cortex, receive probes will be placed 2 to 4 cm from the emitted probe so that they are placed slightly behind C3 or C4 point. The occipital region receive probe will be attached 2 to 4 cm from the emitted probe.
Change of the activation in the somatosensory cortical areas following the noxious stimulation | Measured during painful procedure
  In this study pain will be assessed measuring changes cortical hemodynamics by near-infrared spectroscopy (NIRS). A 2-channel NIRS will be used. The emitted probe provides near-infrared light through on optical fiber will be is placed slightly posterior to Cz position with reference to the international EEG 10-20 system. The receive probes will be fastened over somatosensory and occipital area. In the area of the somatosensory cortex, receive probes will be placed 2 to 4 cm from the emitted probe so that they are placed slightly behind C3 or C4 point. The occipital region receive probe will be attached 2 to 4 cm from the emitted probe.
Change of the activation in the somatosensory cortical areas following the noxious stimulation | Measured immediately after painful procedure
  In this study pain will be assessed measuring changes cortical hemodynamics by near-infrared spectroscopy (NIRS). A 2-channel NIRS will be used. The emitted probe provides near-infrared light through on optical fiber will be is placed slightly posterior to Cz position with reference to the international EEG 10-20 system. The receive probes will be fastened over somatosensory and occipital area. In the area of the somatosensory cortex, receive probes will be placed 2 to 4 cm from the emitted probe so that they are placed slightly behind C3 or C4 point. The occipital region receive probe will be attached 2 to 4 cm from the emitted probe.
Change in heart rate (HR) | Baseline 1, measured pre-intervention
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in heart rate using bedside patient monitor.
Change in heart rate (HR) | Baseline 2, measured pre-procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in heart rate using bedside patient monitor.
Change in heart rate (HR) | Measured during painful procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in heart rate using bedside patient monitor.
Change in heart rate (HR) | Measured immediately after procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in heart rate using bedside patient monitor.
Change in oxygen saturation | Baseline 1, measured pre-intervention
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in oxygen saturation using bedside patient monitor.
Change in oxygen saturation | Baseline 2, measured pre-procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in oxygen saturation using bedside patient monitor.
Change in oxygen saturation | Measured during painful procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in oxygen saturation using bedside patient monitor.
Change in oxygen saturation | Measured immediately after painful procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in oxygen saturation using bedside patient monitor.
Change in respiratory rate | Baseline 1, measured pre-intervention
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in respiratory rate using bedside patient monitor.
Change in respiratory rate | Baseline 2, measured pre-procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in respiratory rate using bedside patient monitor.
Change in respiratory rate | Measured during procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in respiratory rate using bedside patient monitor.
Change in respiratory rate | Measured immediately after procedure
  Neonates' physiological reactions to procedural pain during heel lance will be monitored continuously and measured by recording changes in respiratory rate using bedside patient monitor.

SECONDARY OUTCOMES:
Recovery measured by change in scores of the Premature Infant Pain profile-Revised (PIPP-R) | 3 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the neonates' PIPP-R scores returns to baseline values.
Recovery measured by change in scores of the Premature Infant Pain profile-Revised (PIPP-R) | 5 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the neonates' PIPP-R scores returns to baseline values.
Recovery measured by change in scores of the Premature Infant Pain profile-Revised (PIPP-R) | 10 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the neonates' PIPP-R scores returns to baseline values.
Recovery measured by change in scores of the Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | 3 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the neonates' NIAPAS scores returns to baseline values.
Recovery measured by change in scores of the Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | 5 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the neonates' NIAPAS scores returns to baseline values.
Recovery measured by change in scores of the Neonatal Infant Acute Pain Assessment Scale (NIAPAS) | 10 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the neonates' NIAPAS scores returns to baseline values.
Recovery as measured by changes in somatosensory cortex activation | 3 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the activation in the somatosensory cortical area measured by NIRS returns to baseline values.
Recovery as measured by changes in somatosensory cortex activation | 5 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the activation in the somatosensory cortical area measured by NIRS returns to baseline values.
Recovery as measured by changes in somatosensory cortex activation | 10 minutes after painful procedure
  Time to recovery from painful stimulus will be considered the amount of time in minutes that pass until the activation in the somatosensory cortical area measured by NIRS returns to baseline values
Recovery as measured by changes in heart rate (HR) | 3 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in respiratory rate using a patient monitor.
Recovery as measured by changes in heart rate (HR) | 5 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in respiratory rate using a patient monitor.
Recovery as measured by changes in heart rate (HR) | 10 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in respiratory rate using a patient monitor.
Recovery as measured by changes in oxygen saturation | 3 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in oxygen saturation using a patient monitor.
Recovery as measured by changes in oxygen saturation | 5 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in oxygen saturation using a patient monitor.
Recovery as measured by changes in oxygen saturation | 10 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in oxygen saturation using a patient monitor.
Recovery as measured by changes in respiratory rate | 3 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in respiratory rate using a patient monitor.
Recovery as measured by changes in respiratory rate | 5 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in respiratory rate using a patient monitor.
Recovery as measured by changes in respiratory rate | 10 minutes after painful procedure
  The physiological responses of neonates to recovery from the pain of the procedure are continuously monitored and measured by recording changes in respiratory rate using a patient monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospita, Oulu, Finland